CLINICAL TRIAL: NCT01483807
Title: Treatments of Acquired Apraxia of Speech
Acronym: Apraxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C7419-R
Record Dates: First submitted 2011-04-15; First posted 2011-12-01 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Aphasia; Apraxia of Speech; Stroke
Keywords: speech; speech therapy; apraxia of speech
MeSH Terms: conditions — Aphasia; Apraxias; Stroke; Speech; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Each participant received each arm of treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPT-B then SPT-R (Experimental): Participants first received Sound Production Treatment - Blocked (SPT-B) for 20 treatment sessions spanning approximately 7 weeks. After a washout period of 2 weeks, they then received Sound Production Treatment - Random (SPT-R) for 20 treatment sessions. Follow-up measures were conducted at 2, 6, and 10 weeks following the end of all treatment.
  Interventions: Behavioral: Sound Production Treatment - Blocked; Behavioral: Sound Production Treatment - Random
- SPT-R then SPT-B (Experimental): Participants first received Sound Production Treatment - Random (SPT-R) for 20 treatment sessions spanning approximately 7 weeks. After a washout period of 2 weeks, they then received Sound Production Treatment - Blocked (SPT-B) for 20 treatment sessions. Follow-up measures were conducted at 2, 6, and 10 weeks following the end of all treatment.
  Interventions: Behavioral: Sound Production Treatment - Blocked; Behavioral: Sound Production Treatment - Random

INTERVENTIONS:
Behavioral: Sound Production Treatment - Blocked — Sound Production Treatment is a treatment for acquired apraxia of speech. Combines therapist modeling, simultaneous production, articulatory instruction, feedback and repeated practice. SPT-Blocked entailed practicing all treatment targets blocked by target. SPT-Random entailed practicing all treatment targets in a non predictable, random order.
Behavioral: Sound Production Treatment - Random — A treatment for acquired apraxia of speech. Combines therapist modeling, simultaneous production, articulatory instruction, feedback and repeated practice. SPT-Random entailed practicing treatment targets in a non predictable order. SPT-Blocked entailed practicing treatment targets blocked by target.

SUMMARY:
This study was designed to examine the effects of speech therapy on ability to produce speech sounds in persons with acquired apraxia of speech.

DETAILED DESCRIPTION:
This study was designed to investigate the effects of Sound Production Treatment (SPT; a treatment for acquired apraxia of speech) on sound production accuracy in persons with chronic apraxia of speech (AOS). Organization of practice (blocked practice or randomized practice) will be manipulated in an effort to determine the most efficacious application of SPT. A combination of group and single-subject experimental designs wasl be completed with 20 speakers with AOS (2 groups of 10 participants).

ELIGIBILITY:
Inclusion Criteria:

* Must have acquired apraxia of speech that occurred following a stroke or other brain injury.
* Must be at least 6 months post-onset of brain injury.
* May have aphasia.

Exclusion Criteria:

* History of drug or alcohol abuse.
* History of mental illness.
* Neurological condition other than that which resulted in apraxia of speech.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Wambaugh, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wambaugh JL, Nessler C, Cameron R, Mauszycki SC. Treatment for acquired apraxia of speech: examination of treatment intensity and practice schedule. Am J Speech Lang Pathol. 2013 Feb;22(1):84-102. doi: 10.1044/1058-0360(2012/12-0025). Epub 2012 Oct 15. PMID 23071199
- [Result] Wambaugh J, Shuster L, Bailey DJ, Mauszycki S, Kean J, Nessler C, Wright S, Brunsvold J. Self-Judgments of Word Production Accuracy in Acquired Apraxia of Speech. Am J Speech Lang Pathol. 2016 Dec 1;25(4S):S716-S728. doi: 10.1044/2016_AJSLP-15-0139. PMID 27997948
- [Result] Bailey DJ, Eatchel K, Wambaugh J. Sound Production Treatment: Synthesis and Quantification of Outcomes. Am J Speech Lang Pathol. 2015 Nov;24(4):S798-814. doi: 10.1044/2015_AJSLP-14-0127. PMID 26133692
- [Result] Wambaugh JL, Nessler C, Wright S, Mauszycki SC, DeLong C, Berggren K, Bailey DJ. Effects of Blocked and Random Practice Schedule on Outcomes of Sound Production Treatment for Acquired Apraxia of Speech: Results of a Group Investigation. J Speech Lang Hear Res. 2017 Jun 22;60(6S):1739-1751. doi: 10.1044/2017_JSLHR-S-16-0249. PMID 28655045
- [Result] Mauszycki SC, Bailey DJ, Wambaugh JL. Acquired Apraxia of Speech: The Relationship Between Awareness of Errors in Word Productions and Treatment Outcomes. Am J Speech Lang Pathol. 2017 Jun 22;26(2S):664-673. doi: 10.1044/2017_AJSLP-16-0111. PMID 28654947
- [Result] Wambaugh J, Nessler C, Wright S, Mauszycki S, DeLong C. Sound production treatment for acquired apraxia of speech: Effects of blocked and random practice on multisyllabic word production. Int J Speech Lang Pathol. 2016 Oct;18(5):450-64. doi: 10.3109/17549507.2015.1101161. Epub 2015 Nov 9. PMID 27063676
- [Result] Wambaugh JL, Nessler C, Wright S, Mauszycki SC. Sound production treatment: effects of blocked and random practice. Am J Speech Lang Pathol. 2014 May;23(2):S225-45. doi: 10.1044/2014_AJSLP-13-0072. PMID 24687207
- [Derived] DeLong C, Nessler C, Wright S, Wambaugh J. Semantic Feature Analysis: Further Examination of Outcomes. Am J Speech Lang Pathol. 2015 Nov;24(4):S864-79. doi: 10.1044/2015_AJSLP-14-0155. PMID 26384102

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant received each treatment arm in this cross-over design. Order of treatment assignment was random.
Groups:
- SPT-B Then SPT-R: Participants in this arm received Sound Production Treatment - Blocked (SPT-B) for 20 treatment sessions. Following a 2 week washout period, participants received Sound Production Treatment - Random (SPT-R) for 20 treatment sessions. SPT is a behavioral treatment that includes clinician modeling, orthographic cueing, integral stimulation ("watch me, listen to me, say it with me", articulation instruction, repeated practice and feedback. In the Blocked version, treatment targets are practiced by blocking items by sound target - words with the same target are grouped together. In the Random version, treatment targets are practiced in a non predictable order.
- SPT-R Then SPT-B: Participants in this arm received Sound Production Treatment - Random (SPT-R) for 20 treatment sessions. Following a 2 week washout period, participants received Sound Production Treatment - Blocked (SPT-B) for 20 treatment sessions. SPT is a behavioral treatment that includes clinician modeling, orthographic cueing, integral stimulation ("watch me, listen to me, say it with me", articulation instruction, repeated practice and feedback. In the Blocked version, treatment targets are practiced by blocking items by sound target - words with the same target are grouped together. In the Random version, treatment targets are practiced in a non predictable order.
Period: First Treatment Phase (7 Weeks)
Arm/Group | SPT-B Then SPT-R | SPT-R Then SPT-B
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | SPT-B Then SPT-R | SPT-R Then SPT-B
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Treatment Phase (7 Weeks)
Arm/Group | SPT-B Then SPT-R | SPT-R Then SPT-B
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants received Sound Production Treatment (SPT). Half the participants received SPT applied in a blocked fashion (SPT-B) first for 20 sessions. Following a 2 week washout period, those participants then received SPT applied in random fashion (SPT-R) for 20 sessions. The other half of the participants received the treatments in the opposite order.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/non hispanic | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Accuracy of Articulation [Count of Participants; unit: Participants] — Number of participants with baseline articulation accuracy < 50% correct
  Participants | 20

OUTCOME MEASURES:

1. Primary Outcome: Speech Production: Effect Size for Treated Items
Description: Change in accuracy of articulation of trained items as measured from baseline to 10 weeks post treatment using effect size calculations as the indicator of magnitude of change; production of words designated for treatment was measured repeatedly in non treatment probes prior to treatment, throughout all study phases, and at 10 weeks post treatment with percent accuracy calculated for each probe (maximum = 100%, minimum = 0% correct). Effect size calculations involved calculating the difference between post- and pre-treatment probe accuracy percentages with corrections made for variability (standard deviations in performance). The larger the effect size, the greater the change in performance from pre-treatment. Positive effect sizes = increases in accuracy & negative effect sizes = decreases in accuracy.
Time Frame: Pre treatment (2-3 week period preceding the start of treatment) vs. 10 weeks post all treatment
Population: 20 speakers with chronic apraxia of speech and aphasia; effect sizes were calculated for each speaker for each treatment condition.
Measure: Mean (Full Range); unit: effect size
Groups:
- SPT-R: All Participants: All participants received Sound Production Treatment (SPT). Half the participants received SPT applied in a blocked fashion (SPT-B) first for 20 sessions. Following a 2 week washout period, those participants then received SPT applied in random fashion (SPT-R) for 20 sessions. The other half of the participants received the treatments in the opposite order.All 20 administrations of SPT-R were analyzed relative to all 20 administrations of SPT-B.
- SPT-B: All Participants: All 20 participants received both SPT-R and SPT-B, with order of administration of treatments being counterbalanced across participants. Data for SPT-B are shown here for all of the 20 participants.
Arm/Group | SPT-R: All Participants | SPT-B: All Participants
Number analyzed (Participants) | 20 | 20
effect size | 6.84 [1.66 to 18.78] | 6.14 [.83 to 14.38]
Statistical Analysis 1: Comparison: SPT-R: All Participants vs SPT-B: All Participants; Comparison of performance (change in articulation accuracy) with SPT-R versus SPT-B items. Based on the existing literature, it was predicted that the mean effect size associated with SPT-R would be greater than that for SPT-B; Test type: Superiority; p = .254, t-test, 1 sided; Mean Difference (Final Values) = .70

2. Primary Outcome: Speech Production: Percent Change in Treated Items
Description: Change in accuracy of articulation of treated items as measured by percent increase in accuracy above the highest baseline measurement; production of words designated for treatment was measured repeatedly in non treatment probes prior to treatment, throughout all study phases, and at 10 weeks post treatment with percent accuracy calculated for each probe (0% to 100% correct). The highest percentage accuracy achieved in pre-treatment probes was subtracted from the percentage accuracy achieved at 10 weeks post-treatment to obtain change in accuracy value - this reflects change from maximum correct performance in baseline (pre-treatment). e.g., if in baseline probes, performance ranged from 10% to 30% accuracy and at post treatment performance was 90% accuracy, the change value would be 60% (90% minus 30%). A greater change value indicates greater change in articulation/production of words. Change could be positive (improved articulation) or negative (poorer articulation).
Time Frame: baseline to 10 weeks post treatment
Population: 20 speakers with chronic apraxia of speech and aphasia received both arms of treatment.
Measure: Mean (Full Range); unit: % change
Groups:
- SPT-B: All Participants: All participants received SPT-R and SPT-B with order of treatments counterbalanced. Response to SPT-B is shown here.
Arm/Group | SPT-R: All Participants | SPT-B: All Participants
Number analyzed (Participants) | 20 | 20
% change | 46 [-20 to 100] | 38 [-20 to 80]
Statistical Analysis 1: Comparison: SPT-R: All Participants vs SPT-B: All Participants; On the basis of existing literature. SPT-R was predicted to be associated with greater increase in articulatory accuracy over baseline levels than SPT-B; Test type: Superiority; p = .043, t-test, 1 sided; Mean Difference (Final Values) = 8.25

3. Secondary Outcome: Speech Production: Percent Change in Untrained Items
Description: Percent change in articulatory accuracy of untrained items measured by change in percent accuracy over highest baseline value; production of words designated to NOT receive treatment (untrained items) was measured repeatedly in non treatment probes prior to treatment, throughout all study phases, and at 10 weeks post treatment with percent accuracy calculated for each probe (maximum = 100%, minimum = 0% correct). Effect size calculations involved calculating the difference between post- and pre-treatment probe accuracy percentages with corrections made for variability (standard deviations in performance). The larger the effect size, the greater the change in performance from pre-treatment. Positive effect sizes = increases in accuracy & negative effect sizes = decreases in accuracy.
Time Frame: baseline to 10 weeks post treatment
Population: 20 participants with chronic apraxia of speech and aphasia
Measure: Mean (Full Range); unit: % change
Groups:
- SPT-B: All Participants: All participants received both SPT-R and SPT-B with order of treatments counterbalanced. Results for SPT-B are shown here.
Arm/Group | SPT-R: All Participants | SPT-B: All Participants
Number analyzed (Participants) | 20 | 20
% change | 14 [-60 to 100] | 13 [-60 to 80]
Statistical Analysis 1: Comparison: SPT-R: All Participants vs SPT-B: All Participants; Comparison of change in accuracy of articulation of untreated items: SPT-R versus SPT-B items. It was predicted that there would be a greater increase in accuracy for SPT-R items; Test type: Superiority; p = .396, t-test, 1 sided

4. Secondary Outcome: Speech Production of Untrained Items: Effect Sizes for Untrained Items
Description: Change in accuracy of articulation of untrained items as measured by effect sizes reflecting magnitude of change. Production of words designated to not receive treatment (i.e., generalization items) was measured repeatedly in non treatment probes prior to treatment, throughout all study phases, and at 10 weeks post treatment with percent accuracy calculated for each probe (0% to 100% correct). Change in accuracy of articulation of untrained items was measured from baseline to 10 weeks post treatment using effect size calculations as the indicator of magnitude of change. Effect size calculations involved calculating the difference between post- and pre-treatment probe accuracy percentages with corrections made for variability (standard deviations in performance). The larger the effect size, the greater the change in performance from pre-treatment.
Time Frame: Baseline vs. 10 weeks post all treatment
Population: 20 speakers with chronic apraxia of speech and aphasia
Measure: Mean (Full Range); unit: effect size
Groups:
- SPT-B: All Participants: All participants received both SPT-R and SPT-B with order of treatments counterbalanced. SPT-B results are shown here.
Arm/Group | SPT-R: All Participants | SPT-B: All Participants
Number analyzed (Participants) | 20 | 20
effect size | 2.56 [-.29 to 9.84] | 2.11 [-.77 to 7.83]
Statistical Analysis 1: Comparison: SPT-R: All Participants vs SPT-B: All Participants; Comparison of effect sizes obtained for untreated SPT-R versus untreated SPT-B items. It was predicted that effect sizes would be greater for SPT-R untreated items; Test type: Superiority; p = .212, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Entire course of study which was approximately 30 weeks per participant: pretreatment/baseline period = 4 weeks + 7 weeks Treatment 1 + 2 weeks washout + 7 weeks Treatment 2 + follow-up at 10 weeks.
Groups:
- All Participants: All participants received Sound Production Treatment (SPT). Half of the participants received SPT administered in a blocked fashion (SPT-B) first, followed by a 2 week washout period, and then SPT administered in a random fashion (SPT-R). The other half of the participants received both treatments administered in the reverse order. Participants were grouped together for analyses by treatment type; this was due to the fact that all participants received both treatments and were observed in the same way for both treatments regardless of which treatment was received first. There were not adverse events and consequently, no need to examine adverse events by arm.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Two participants, one in each arm, received 10 sessions per phase rather than 20 sessions. This was due to these participants achieving high levels of accuracy very quickly; 20 sessions were not required (reduced burden).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2015-11-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT01483807/Prot_000.pdf
  • Informed Consent Form (2015-11-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT01483807/ICF_001.pdf
  • Statistical Analysis Plan (2015-11-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT01483807/SAP_002.pdf